CLINICAL TRIAL: NCT00625040
Title: Incretin Physiology and Beta-cell Function Before and After Weight-loss - Effects of Long-term Weight Loss Following Laparoscopic Adjustable Gastric Banding
Brief Title: Incretin Physiology and Beta-cell Function Before and After Weight-loss
Status: Terminated | Type: Observational
Why Stopped: Not enough patients in the follow-up period
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: University of Copenhagen (Other); European Foundation for the Study of Diabetes (Other); Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Katrine Bagge Hansen, MD, Ph.d, Glostrup University Hospital, Copenhagen
Other Study IDs: GB-INK
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Obesity
Keywords: Incretin effect; Gastric banding; Glucagon; Glucagon-Like Peptide 1; Gastric Inhibitory Peptide; Glucose Intestinal Peptide; Insulin; C-peptide
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — p-glucose, p-glucagon, p-GLP1, p-GIP, p-cpeptid, p-insulin, p-paracetamol, buffy coat, urine, whole blood sampels
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A: Obese patients without diabetes with a Body Mass Index > 37 kg/m2
  Interventions: Other: Oral glucose tolerance test (OGTT), isoglycemic iv. clamp, liquid meal test, gastric emptying rate

INTERVENTIONS:
Other: Oral glucose tolerance test (OGTT), isoglycemic iv. clamp, liquid meal test, gastric emptying rate — OGTT: The test is performed with 50 g of glucose deluded in 300 ml water
  Isoglycemic iv. clamp: Iv. glucose infusion mimicking the glucose response curves from the OGTT
  Liquid Meal test: The test is performed with 100g of formula milk deluded in 300 ml. water
  Gastric Emptying Rate: Paracetamol absorption test.

SUMMARY:
To evaluate the impact of laparoscopic adjustable gastric banding (LAGB) on beta-cell function, insulin sensitivity, incretin function, postprandial secretion of incretin hormones (glucagon-like peptide-1 (GLP-1) and glucose-dependent insulinotropic polypeptide (GIP)) in morbidly obese patients and to describe the pathophysiological mechanisms involved in the amelioration of glucose homeostasis during long-term weight loss.

DETAILED DESCRIPTION:
Morbid obesity represents a serious health issue in Western countries, with a rising incidence and a strong association with increased mortality and serious co-morbidities, such as diabetes. Surgical interventions, such as laparoscopic gastric banding have been developed with the aim of providing a laparoscopic placed device that is safe and effective in generating substantial weight loss. By investigation of the incretin effect, the secretion of GIP and GLP-1, the insulin response and sensitivity and the beta-cell responsiveness to glucose in 10 obese patients without type 2 diabetes before and after laparoscopic gastric banding the aim of this project is describe the pathophysiological mechanisms involved in the amelioration of glucose homeostasis during long-term weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Caucasians without type 2 diabetes mellitus
* Normal OGTT (75 g of glucose) according to WHO's criteria
* Patients fulfilling the criteria for laparoscopic gastric banding
* Normal Hemoglobin
* Informed consent

Exclusion Criteria:

* Liver disease (ALAT > 2 x normal level)
* Nephropathy (s-creatinin > 130 µM or albuminuria)
* Relatives (parents/siblings) with T2DM
* Medical treatment witch cannot be stopped for 12 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cases and controls are recruited from The Bariatric Clinic at Glostrup Hospital
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2008-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Incretin effect before and one year after gastric banding in obese patients without diabetes | One year

SECONDARY OUTCOMES:
GLP-1 and GIP response curves | One year

CONTACTS AND LOCATIONS:
Overall Officials: Katrine Bagge Hansen, MD, Principal Investigator — Glostrup University Hospital, Copenhagen; Filip K Knop, MD, PhD, Study Director — Gentofte Hospital; Steen Larsen, MD, DMSc, Study Director — Glostrup University Hospital, Copenhagen; Jens Juul Holst, MD,DMSc, Study Director — University of Copenhagen; Viggo Kristensen, MD, Study Chair — Glostrup University Hospital, Copenhagen
Locations (1):
- Glostrup Hospital, Glostrup Municipality, Denmark